CLINICAL TRIAL: NCT06592209
Title: Body Electric: a Pragmatic Trial Evaluating Movement Breaks As a Public Health Strategy to Mitigate the Harms of Prolonged Sedentary Behavior
Brief Title: Body Electric: a Pragmatic Trial Evaluating the Viability of Movement Breaks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Keith Diaz, Associate Professor of Behavioral Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAU8061
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sedentary Behavior
Keywords: Sedentary Behavior; Fatigue; Mood; Work Performance; Work Engagement; Implementation; Barriers; Intervention; Movement Breaks; Facilitators
MeSH Terms: conditions — Sedentary Behavior; Fatigue

STUDY DESIGN:
Intervention Model Description: Three-arm trial wherein participants self-selected a movement break dose to follow (5 min movement breaks every 30, 60, or 120 min)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Every 30 Minutes Movement Break (Experimental): Participants in the movement breaks every 30 minutes group complete a 7-day baseline period, followed by 2 weeks of the selected dose condition. Participants are asked to complete movement breaks every 30 minutes during all waking hours on weekdays and weekends (i.e. 7 days a week). Information regarding work productivity, energy and fatigue levels, mood, physical activity, and barriers/facilitators to taking movement breaks are collected via either 5 daily SMS surveys throughout the day (9am, 12pm, 3pm, 6pm, 9pm) or one emailed survey at the end of each day (8pm). Survey delivery method is randomized. Participants also provide feedback regarding the feasibility, acceptability, and appropriateness of the intervention.
  Interventions: Behavioral: Sedentary Breaks
- Every 60 Minutes Movement Break (Experimental): Participants in the movement breaks every 60 minutes group complete a 7-day baseline period, followed by 2 weeks of the selected dose condition. Participants are asked to complete movement breaks every 60 minutes during all waking hours on weekdays and weekends (i.e. 7 days a week). Information regarding work productivity, energy and fatigue levels, mood, physical activity, and barriers/facilitators to taking movement breaks are collected via either 5 daily SMS surveys throughout the day (9am, 12pm, 3pm, 6pm, 9pm) or one emailed survey at the end of each day (8pm). Survey delivery method is randomized. Participants also provide feedback regarding the feasibility, acceptability, and appropriateness of the intervention.
  Interventions: Behavioral: Sedentary Breaks
- Every 120 Minutes Movement Break (Experimental): Participants in the movement breaks every 120 minutes group complete a 7-day baseline period, followed by 2 weeks of the selected dose condition. Participants are asked to complete movement breaks every 120 minutes during all waking hours on weekdays and weekends (i.e. 7 days a week). Information regarding work productivity, energy and fatigue levels, mood, physical activity, and barriers/facilitators to taking movement breaks are collected via either 5 daily SMS surveys throughout the day (9am, 12pm, 3pm, 6pm, 9pm) or one emailed survey at the end of each day (8pm). Survey delivery method is randomized. Participants also provide feedback regarding the feasibility, acceptability, and appropriateness of the intervention.
  Interventions: Behavioral: Sedentary Breaks

INTERVENTIONS:
Behavioral: Sedentary Breaks — Participants recruited through a podcast series (Body Electric) produced by National Public Radio were asked to select one of three movement break conditions (5 minutes of movement for every 30-, 60-, or 120-minutes of sedentary time). Participants are asked to complete movement breaks during all waking hours on weekdays and weekends (i.e. 7 days a week). During movement breaks, participants are instructed to walk for 5 minutes in whichever way was most comfortable and safe (i.e. self-selected pace and location). Participants who use an assistive device such as a wheelchair or walker, were instructed to wheel, walk, or complete other convenient, comfortable, and safe types of movement such as upper body exercises with resistance bands, chair-based exercises, etc. No break reminders were provided, although participants were encouraged to set reminders in their phones or to utilize commercially available apps or wearable devices.
  Other Names: Movement Breaks

SUMMARY:
The purpose of this pragmatic trial is to determine the implementation potential of three movement break doses (every 30, 60, or 90 min) under real-world conditions. The main questions it aims to answer are:

* What is the feasibility, acceptability, appropriateness, and compliance to the tested movement break doses under real-world conditions?
* What is the effectiveness of the movement break doses on improving mood, fatigue, and work performance?
* What are the barriers of and facilitators to taking movement breaks across population subgroups (age group, sex, race/ethnicity, employment status, employment setting, and occupation).

Researchers will compare differences in the primary (implementation metrics), secondary (mood, fatigue, and work performance), and exploratory (barriers/facilitators) outcomes across the three trial arms (movement breaks every 30, 60, or 120 minutes).

Participants will:

* Take movement breaks (5 minutes of walking at a self-selected pace) daily according to their dose condition (every 30, 60, or 90 minutes) for two consecutive weeks.
* Complete daily surveys to report compliance, barriers/facilitators, and mood/fatigue/work performance.
* Complete a survey battery at the end of the study to report implementation potential, rank/rate barriers and facilitators, and evaluate mood/fatigue/work performance.

To address the study aims, the investigator will recruit 50,000 adults and will conduct a dosing study that concurrently tests three movement break doses. Participants will complete a 7-day baseline period to assess normal durations of sedentary behavior and movement, followed by a 2-week period during which they will be select a movement break dose to implement in their everyday life for the duration of the program. The break frequency x duration combination will include 5 minute every 30 minutes, 5 minutes every 60 minutes, and 5 minutes every 120 minutes. Work and leisure behaviors, mood, fatigue, and barriers/facilitators will be assessed via survey at enrollment, as well as via daily surveys during the baseline and intervention monitoring periods.

DETAILED DESCRIPTION:
U.S. adults spend on average ~11-12 h/day sedentary. Accordingly, the phrase "sitting is the new smoking" has been used to describe an epidemic of developed nations. Daily sedentary time is strongly associated with risk for cardiovascular disease (CVD) morbidity and mortality, irrespective of moderate-vigorous physical activity (MVPA). As such, the 2018 Physical Activity Guidelines for Americans, have expanded beyond promoting MVPA and now also advocate for reductions in sedentary time. These recommendations, however, are very general ("sit less, move more") due to a paucity of data to inform more quantitative recommendations. To inform more specific guidelines, both the 2018 Physical Activity Guidelines Advisory Committee Scientific Report and a scientific advisory on sedentary behavior from the American Heart Association (AHA) have identified a critical research need for studies that compare different doses of reducing sedentary time on health outcomes and evaluate the barriers to real-world implementation of sedentary time reduction strategies. Such studies were deemed to be critical for development of evidence based sedentary behavior guidelines. The proposed study will address this major evidence gap and provide evidence to inform the feasibility of specific, quantitative movement break sedentary behavior recommendations.

Research has implicated sedentary time accrued in prolonged, uninterrupted bouts (e.g., sitting for hours at a time) as potentially the most hazardous form of sedentary behavior; suggestive that regularly breaking up sedentary time with bouts of activity may be an important adjunct to existing physical activity guidelines. Although these data inform which sedentary behavior feature to target, they provide little to inform quantitative guidelines. Thus, only general recommendations to "sit less, move more" have been proposed without specific, actionable targets. The investigator's latest laboratory-based research has documented quantitative guidance regarding (1) How frequent should periods of prolonged sedentary time be interrupted? and (2) What is the appropriate duration of these breaks in sedentary time? However, it is unclear how feasible and acceptable these quantitative recommendations (i.e., taking a walking break every half hour for 5 minutes) are. Moreover, the barriers to and facilitators of successfully implementing breaks in sedentary time during the day are largely unknown.

Primary Aim: To determine the feasibility, acceptability, and appropriateness (i.e., the implementation potential) of and compliance to three movement break doses (every 30, 60, or 120 minutes) under real world conditions.

Secondary Aim: To determine the effect of various movement break doses on mood, fatigue, and work performance.

Exploratory Aim: The successful implementation of movement breaks into mainstream society relies on an understanding of common facilitators and barriers to movement breaks faced by the public across a vast array of population subgroups. This study will map barriers to and facilitators of movement breaks by age group (young, middle-aged, and older adults), sex, race/ethnicity, employment status (full-time, part-time, retired, not working), employment setting (remote, in-person, hybrid), and occupation type.

Excessive sedentary time is highly prevalent in developed nations and linked to increased CVD risk. No evidence-based recommendations exist on how people should break up sedentary time. Evaluating the implementation potential of doses (in frequency and duration) of a movement break intervention that yields improvements across several health indices and establishing barriers/facilitators to movement breaks across population subgroups could have a powerful impact on public health by establishing a recommended movement break dose for future randomized trials and guidelines and laying the foundation to optimize future movement break interventions that address population barriers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English speaking
* Access to a smart phone with a data and text messaging plan

Exclusion Criteria:

* Recent history of bone, joint, or soft tissue injury that would be worsened by exercise
* Chest pain at rest, during activities of daily living, or with movement
* Instructions from a physician requiring supervised exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20217 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) Score | 2 weeks
  Feasibility - Measured by the Feasibility of Intervention Measure (FIM) instrument. The FIM is a 4-item survey that measures the extent to which a new treatment, or an intervention, can be successfully used or carried out within a given setting. This is assessed at study completion via an end-of-study survey. Items are rated on a 5-point Likert scale from completely disagree to completely agree. Higher scores reflect higher feasibility of the intervention.
Acceptability of Intervention Measure (AIM) Score | 2 weeks
  Acceptability - Measured by the Acceptability of Intervention Measure (AIM) instrument. The AIM is a 4-item survey that measures the extent to which a new treatment, or an intervention, is agreeable, palatable, or satisfactory. This is assessed at study completion via an end-of-study survey. Items are rated on a 5-point Likert scale from completely disagree to completely agree. Higher scores reflect higher acceptability of the intervention.
Intervention Appropriateness Measures (IAM) Score | 2 weeks
  Appropriateness - Measured by the Intervention Appropriateness Measures (IAM). The IAM is a 4-item survey that measures the perceived fit, relevance, or compatibility of a new treatment, or an intervention, for a given setting or consumer, and/or the perceived fit of the treatment/intervention to address a particular issue or problem. This is assessed at study completion via an end-of-study survey. Items are rated on a 5-point Likert scale from completely disagree to completely agree. Higher scores reflect higher appropriateness of the intervention.
Number of Movement Breaks | 2 weeks
  This is to measure compliance to the movement break condition. Completion of movement breaks is assessed using surveys either delivered via SMS 5 times per day or via one end of day survey (survey delivery method determined randomly). Participants self-report the number and duration of sedentary breaks completed since the last survey.

SECONDARY OUTCOMES:
Fatigue Symptom Inventory (FSI) Score | 2 weeks
  Physical exhaustion and fatigue are assessed using the Fatigue Symptom Inventory-3 (FSI-3). The instrument consists of 3 exhaustion/fatigued-related items ("Average fatigue", "Fatigue interference with activity levels", "Fatigue interference with enjoyment of life") with response options on a 10-point scale from 0 (Not at all fatigued/No interference) to 10 (As fatigued as I could be/Extreme interference). Responses are summed with higher scores indicating greater perceived physical exhaustion/fatigued.
Positive and Negative Affect Schedule (PANAS) Short Form Score | 2 weeks
  Positive and negative affect are measured using the Positive and Negative Affect Schedule (PANAS) Short Form. This instrument contains 10 items wherein participants respond to words (i.e., hostile, nervous, attentive, inspired) that describe different feelings and emotions and indicate the extent they felt this way on a 5-point Likert scale from very slightly or not at all to extremely. The positive and negative affect subscales are each scored with higher scores reflecting higher positive/negative affect.
Work Performance Score | 2 weeks
  Perceived work performance quantity and quality, along with an overall rating of work performance, are measured by the World Health Organization Health and Work Performance Questionnaire (HPQ). The HPQ includes two items that measure performance quantity (e.g., How often did you not work at times when you were supposed to be working;) and three items that measure performance quality on a 5-point Likert scale; along with an overall rating of work performance on a 0 to 10 scale. Higher scores reflect higher perceived work performance.
Utrecht Work Engagement Scale (UWES-3) Score | 2 weeks
  Work engagement is assessed using a shortened-version of the Utrecht Work Engagement Scale (UWES-3). It is composed of three items wherein participants rate the extent to which they experienced feelings of energy, enthusiasm, and immersion during work on a 7-point scale from never to always. Higher scores reflect higher work engagement.
Fatigue Visual Analog Scale (VAS) Score | 2 weeks
  Momentary or daily fatigued are assessed with a single item (i.e., How fatigued are you right now? How fatigued were you today?) on a visual analogue scale (VAS) from 0 (anchor: no fatigue at all) to 100 (anchor: extremely fatigued). A slider that moved in 1-point increments is used to indicate responses. Single item fatigue VAS scores are assessed using surveys either delivered via SMS 5 times per day (momentary assessments) or via one end of day survey (daily assessment). Survey delivery method is determined randomly.
Affect Visual Analog Scale (VAS) Score | 2 weeks
  Momentary or daily affect is assessed with a single item (i.e., how do you feel right now? How did you feel today?) on a visual analogue scale (VAS) from -50 (anchor: very negative) to +50 (anchor: very positive). A slider that moves in 1-point increments is used to indicate responses. Single item affect VAS scores are assessed using surveys either delivered via SMS 5 times per day (momentary assessments) or via one end of day survey (daily assessment). Survey delivery method is determined randomly.
Work Performance Visual Analog Scale (VAS) Score | 2 weeks
  Daily work performance is assessed with a single item (how would you rate your overall job performance today?) on a visual analogue scale (VAS) from 0 (anchor: worst performance) to 10 (anchor: top performance). A slider that moves in 1-point increments is used to indicate responses.

OTHER OUTCOMES:
Percentage of participants that experienced barriers to movement break completion | 2-week intervention period
  This measure assesses the challenges (barriers) that participants face that inhibit them from completing movement breaks. During the intervention period, barriers are assessed using surveys either delivered via SMS 5 times per day or via one end of day survey (survey delivery method determined randomly). Participants are asked to select from a list of 18 common barriers or report via open text response other barriers not listed that they faced since the last survey. During the end-of-study survey, participants also rate the extent to which they experienced each barrier on 5-point Likert scale and rank their top three barriers.
Sedentary Time | 2 weeks
  Sedentary time is assessed using the Sedentary Behavior Questionnaire (SBQ). The SBQ assesses the amount of time spent doing 9 sedentary behaviors (watching television, playing computer/video games, sitting while listening to music, sitting and talking on the phone, doing paperwork or office work, sitting and reading, playing a musical instrument, doing arts and crafts, sitting and driving/riding in a car, bus, or train). The 9 items are completed separately for weekdays and weekend days. The time reported for each item are summed to derive daily sedentary time values expressed in minutes per day.
Percentage of participants that experienced facilitator to movement break completion | 2 weeks
  This measure assesses the strategies (or facilitators) that participants used to help them complete movement break protocol. During the intervention period, facilitators are assessed using surveys either delivered via SMS 5 times per day or via one end of day survey (survey delivery method determined randomly). Participants are asked to select from a list of 11 common facilitators or report via open text response other facilitators not listed that helped them take a movement break since the last survey. During the end-of-study survey, participants are also asked to rate and rank facilitators. During the end-of-study survey, participants also rate the extent to which they utilized each facilitator on 5-point Likert scale and rank their top three facilitators.

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Diaz, PhD, Principal Investigator — Florence Irving Associate Professor of Behavioral Medicine
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Archer E, Shook RP, Thomas DM, Church TS, Katzmarzyk PT, Hebert JR, McIver KL, Hand GA, Lavie CJ, Blair SN. 45-Year trends in women's use of time and household management energy expenditure. PLoS One. 2013;8(2):e56620. doi: 10.1371/journal.pone.0056620. Epub 2013 Feb 20. PMID 23437187
- [Background] Church TS, Earnest CP, Skinner JS, Blair SN. Effects of different doses of physical activity on cardiorespiratory fitness among sedentary, overweight or obese postmenopausal women with elevated blood pressure: a randomized controlled trial. JAMA. 2007 May 16;297(19):2081-91. doi: 10.1001/jama.297.19.2081. PMID 17507344
- [Background] van der Ploeg HP, Venugopal K, Chau JY, van Poppel MNM, Breedveld K, Merom D, Bauman AE. Non-occupational sedentary behaviors: population changes in The Netherlands, 1975-2005. Am J Prev Med. 2013 Apr;44(4):382-387. doi: 10.1016/j.amepre.2012.11.034. PMID 23498104
- [Background] Dunstan DW, Howard B, Healy GN, Owen N. Too much sitting--a health hazard. Diabetes Res Clin Pract. 2012 Sep;97(3):368-76. doi: 10.1016/j.diabres.2012.05.020. Epub 2012 Jun 9. PMID 22682948
- [Background] Brownson RC, Boehmer TK, Luke DA. Declining rates of physical activity in the United States: what are the contributors? Annu Rev Public Health. 2005;26:421-43. doi: 10.1146/annurev.publhealth.26.021304.144437. PMID 15760296
- [Background] Diaz KM, Howard VJ, Hutto B, Colabianchi N, Vena JE, Blair SN, Hooker SP. Patterns of Sedentary Behavior in US Middle-Age and Older Adults: The REGARDS Study. Med Sci Sports Exerc. 2016 Mar;48(3):430-8. doi: 10.1249/MSS.0000000000000792. PMID 26460633
- [Background] Biswas A, Oh PI, Faulkner GE, Bajaj RR, Silver MA, Mitchell MS, Alter DA. Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Ann Intern Med. 2015 Jan 20;162(2):123-32. doi: 10.7326/M14-1651. PMID 25599350
- [Background] Diaz KM, Howard VJ, Hutto B, Colabianchi N, Vena JE, Safford MM, Blair SN, Hooker SP. Patterns of Sedentary Behavior and Mortality in U.S. Middle-Aged and Older Adults: A National Cohort Study. Ann Intern Med. 2017 Oct 3;167(7):465-475. doi: 10.7326/M17-0212. Epub 2017 Sep 12. PMID 28892811
- [Background] Thorp AA, Owen N, Neuhaus M, Dunstan DW. Sedentary behaviors and subsequent health outcomes in adults a systematic review of longitudinal studies, 1996-2011. Am J Prev Med. 2011 Aug;41(2):207-15. doi: 10.1016/j.amepre.2011.05.004. PMID 21767729
- [Background] Wilmot EG, Edwardson CL, Achana FA, Davies MJ, Gorely T, Gray LJ, Khunti K, Yates T, Biddle SJ. Sedentary time in adults and the association with diabetes, cardiovascular disease and death: systematic review and meta-analysis. Diabetologia. 2012 Nov;55(11):2895-905. doi: 10.1007/s00125-012-2677-z. Epub 2012 Aug 14. PMID 22890825
- [Background] Ekelund U, Tarp J, Steene-Johannessen J, Hansen BH, Jefferis B, Fagerland MW, Whincup P, Diaz KM, Hooker SP, Chernofsky A, Larson MG, Spartano N, Vasan RS, Dohrn IM, Hagstromer M, Edwardson C, Yates T, Shiroma E, Anderssen SA, Lee IM. Dose-response associations between accelerometry measured physical activity and sedentary time and all cause mortality: systematic review and harmonised meta-analysis. BMJ. 2019 Aug 21;366:l4570. doi: 10.1136/bmj.l4570. PMID 31434697
- [Background] Patterson R, McNamara E, Tainio M, de Sa TH, Smith AD, Sharp SJ, Edwards P, Woodcock J, Brage S, Wijndaele K. Sedentary behaviour and risk of all-cause, cardiovascular and cancer mortality, and incident type 2 diabetes: a systematic review and dose response meta-analysis. Eur J Epidemiol. 2018 Sep;33(9):811-829. doi: 10.1007/s10654-018-0380-1. Epub 2018 Mar 28. PMID 29589226
- [Background] Young DR, Hivert MF, Alhassan S, Camhi SM, Ferguson JF, Katzmarzyk PT, Lewis CE, Owen N, Perry CK, Siddique J, Yong CM; Physical Activity Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Functional Genomics and Translational Biology; and Stroke Council. Sedentary Behavior and Cardiovascular Morbidity and Mortality: A Science Advisory From the American Heart Association. Circulation. 2016 Sep 27;134(13):e262-79. doi: 10.1161/CIR.0000000000000440. Epub 2016 Aug 15. PMID 27528691
- [Background] Heron L, O'Neill C, McAneney H, Kee F, Tully MA. Direct healthcare costs of sedentary behaviour in the UK. J Epidemiol Community Health. 2019 Jul;73(7):625-629. doi: 10.1136/jech-2018-211758. Epub 2019 Mar 25. PMID 30910857
- [Background] Katzmarzyk PT, Powell KE, Jakicic JM, Troiano RP, Piercy K, Tennant B; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Sedentary Behavior and Health: Update from the 2018 Physical Activity Guidelines Advisory Committee. Med Sci Sports Exerc. 2019 Jun;51(6):1227-1241. doi: 10.1249/MSS.0000000000001935. PMID 31095080
- [Background] Matthews CE, George SM, Moore SC, Bowles HR, Blair A, Park Y, Troiano RP, Hollenbeck A, Schatzkin A. Amount of time spent in sedentary behaviors and cause-specific mortality in US adults. Am J Clin Nutr. 2012 Feb;95(2):437-45. doi: 10.3945/ajcn.111.019620. Epub 2012 Jan 4. PMID 22218159
- [Background] Saunders TJ, Larouche R, Colley RC, Tremblay MS. Acute sedentary behaviour and markers of cardiometabolic risk: a systematic review of intervention studies. J Nutr Metab. 2012;2012:712435. doi: 10.1155/2012/712435. Epub 2012 Jun 17. PMID 22754695
- [Background] Duvivier BM, Schaper NC, Bremers MA, van Crombrugge G, Menheere PP, Kars M, Savelberg HH. Minimal intensity physical activity (standing and walking) of longer duration improves insulin action and plasma lipids more than shorter periods of moderate to vigorous exercise (cycling) in sedentary subjects when energy expenditure is comparable. PLoS One. 2013;8(2):e55542. doi: 10.1371/journal.pone.0055542. Epub 2013 Feb 13. PMID 23418444
- [Background] Prince SA, Saunders TJ, Gresty K, Reid RD. A comparison of the effectiveness of physical activity and sedentary behaviour interventions in reducing sedentary time in adults: a systematic review and meta-analysis of controlled trials. Obes Rev. 2014 Nov;15(11):905-19. doi: 10.1111/obr.12215. Epub 2014 Aug 11. PMID 25112481
- [Background] Piercy KL, Troiano RP, Ballard RM, Carlson SA, Fulton JE, Galuska DA, George SM, Olson RD. The Physical Activity Guidelines for Americans. JAMA. 2018 Nov 20;320(19):2020-2028. doi: 10.1001/jama.2018.14854. PMID 30418471
- [Background] Davies S, Atherton F, McBride M, Calderwood C. UK Chief Medical Officers' Physical Activity Guidelines. Chief Medical Officers. 2019.
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Background] Zealand N, McIntyre L, Dutton M. Eating and activity guidelines for new zealand adults. Ministry of Health; 2015.
- [Background] Australian Government Department of Health. Australia's physical activity and sedentary behaviour guidelines. Dep Heal Website. 2014.
- [Background] Tremblay MS, Carson V, Chaput JP, Connor Gorber S, Dinh T, Duggan M, Faulkner G, Gray CE, Gruber R, Janson K, Janssen I, Katzmarzyk PT, Kho ME, Latimer-Cheung AE, LeBlanc C, Okely AD, Olds T, Pate RR, Phillips A, Poitras VJ, Rodenburg S, Sampson M, Saunders TJ, Stone JA, Stratton G, Weiss SK, Zehr L. Canadian 24-Hour Movement Guidelines for Children and Youth: An Integration of Physical Activity, Sedentary Behaviour, and Sleep. Appl Physiol Nutr Metab. 2016 Jun;41(6 Suppl 3):S311-27. doi: 10.1139/apnm-2016-0151. PMID 27306437
- [Background] Fuzeki E, Vogt L, Banzer W. [German National Physical Activity Recommendations for Adults and Older Adults: Methods, Database and Rationale]. Gesundheitswesen. 2017 Mar;79(S 01):S20-S28. doi: 10.1055/s-0042-123700. Epub 2017 Apr 11. German. PMID 28399582
- [Background] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Background] Physical Activity Guidelines Advistory Committee. Physical activity guidelines advisory committee report, 2018. Washington, DC: US Department of Health and Human Services; 2018.
- [Background] Chastin SF, Egerton T, Leask C, Stamatakis E. Meta-analysis of the relationship between breaks in sedentary behavior and cardiometabolic health. Obesity (Silver Spring). 2015 Sep;23(9):1800-10. doi: 10.1002/oby.21180. PMID 26308477
- [Background] Saunders TJ, Atkinson HF, Burr J, MacEwen B, Skeaff CM, Peddie MC. The Acute Metabolic and Vascular Impact of Interrupting Prolonged Sitting: A Systematic Review and Meta-Analysis. Sports Med. 2018 Oct;48(10):2347-2366. doi: 10.1007/s40279-018-0963-8. PMID 30078066
- [Background] Dunstan DW, Kingwell BA, Larsen R, Healy GN, Cerin E, Hamilton MT, Shaw JE, Bertovic DA, Zimmet PZ, Salmon J, Owen N. Breaking up prolonged sitting reduces postprandial glucose and insulin responses. Diabetes Care. 2012 May;35(5):976-83. doi: 10.2337/dc11-1931. Epub 2012 Feb 28. PMID 22374636
- [Background] Howard BJ, Fraser SF, Sethi P, Cerin E, Hamilton MT, Owen N, Dunstan DW, Kingwell BA. Impact on hemostatic parameters of interrupting sitting with intermittent activity. Med Sci Sports Exerc. 2013 Jul;45(7):1285-91. doi: 10.1249/MSS.0b013e318285f57e. PMID 23439415
- [Background] Bailey DP, Locke CD. Breaking up prolonged sitting with light-intensity walking improves postprandial glycemia, but breaking up sitting with standing does not. J Sci Med Sport. 2015 May;18(3):294-8. doi: 10.1016/j.jsams.2014.03.008. Epub 2014 Mar 20. PMID 24704421
- [Background] Carter SE, Draijer R, Holder SM, Brown L, Thijssen DHJ, Hopkins ND. Effect of different walking break strategies on superficial femoral artery endothelial function. Physiol Rep. 2019 Aug;7(16):e14190. doi: 10.14814/phy2.14190. PMID 31423757
- [Background] Scutti S. Yes, sitting too long can kill you, even if you exercise. CNN. 2017
- [Background] Peddie MC, Bone JL, Rehrer NJ, Skeaff CM, Gray AR, Perry TL. Breaking prolonged sitting reduces postprandial glycemia in healthy, normal-weight adults: a randomized crossover trial. Am J Clin Nutr. 2013 Aug;98(2):358-66. doi: 10.3945/ajcn.112.051763. Epub 2013 Jun 26. PMID 23803893
- [Background] Altenburg TM, Rotteveel J, Dunstan DW, Salmon J, Chinapaw MJ. The effect of interrupting prolonged sitting time with short, hourly, moderate-intensity cycling bouts on cardiometabolic risk factors in healthy, young adults. J Appl Physiol (1985). 2013 Dec;115(12):1751-6. doi: 10.1152/japplphysiol.00662.2013. Epub 2013 Oct 17. PMID 24136111
- [Background] Czajkowski SM. News from NIH: using basic behavioral science to develop better behavioral interventions. Transl Behav Med. 2011 Dec;1(4):507-8. doi: 10.1007/s13142-011-0079-2. No abstract available. PMID 24073070
- [Background] Czajkowski SM, Powell LH, Adler N, Naar-King S, Reynolds KD, Hunter CM, Laraia B, Olster DH, Perna FM, Peterson JC, Epel E, Boyington JE, Charlson ME. From ideas to efficacy: The ORBIT model for developing behavioral treatments for chronic diseases. Health Psychol. 2015 Oct;34(10):971-82. doi: 10.1037/hea0000161. Epub 2015 Feb 2. PMID 25642841
- [Background] Naar S, Czajkowski SM, Spring B. Innovative study designs and methods for optimizing and implementing behavioral interventions to improve health. Health Psychol. 2018 Dec;37(12):1081-1091. doi: 10.1037/hea0000657. Epub 2018 Oct 11. PMID 30307270
- [Background] National Institute of Aging. The NIH Stage Model for behavioral intervention development. https://www.nia.nih.gov/research/dbsr/nih-stage-model-behavioral-intervention-development.
- [Background] Prince SA, Reed JL, Cotie LM, Harris J, Pipe AL, Reid RD. Results of the Sedentary Intervention Trial in Cardiac Rehabilitation (SIT-CR Study): A pilot randomized controlled trial. Int J Cardiol. 2018 Oct 15;269:317-324. doi: 10.1016/j.ijcard.2018.07.082. Epub 2018 Jul 19. PMID 30072156
- [Background] Elkind MS, Sacco RL, MacArthur RB, Fink DJ, Peerschke E, Andrews H, Neils G, Stillman J, Corporan T, Leifer D, Cheung K. The Neuroprotection with Statin Therapy for Acute Recovery Trial (NeuSTART): an adaptive design phase I dose-escalation study of high-dose lovastatin in acute ischemic stroke. Int J Stroke. 2008 Aug;3(3):210-8. doi: 10.1111/j.1747-4949.2008.00200.x. PMID 18705902
- [Background] Muler JH, McGinn CJ, Normolle D, Lawrence T, Brown D, Hejna G, Zalupski MM. Phase I trial using a time-to-event continual reassessment strategy for dose escalation of cisplatin combined with gemcitabine and radiation therapy in pancreatic cancer. J Clin Oncol. 2004 Jan 15;22(2):238-43. doi: 10.1200/JCO.2004.03.129. Epub 2003 Dec 9. PMID 14665608
- [Background] Gordon PH, Cheung YK, Levin B, Andrews H, Doorish C, Macarthur RB, Montes J, Bednarz K, Florence J, Rowin J, Boylan K, Mozaffar T, Tandan R, Mitsumoto H, Kelvin EA, Chapin J, Bedlack R, Rivner M, McCluskey LF, Pestronk A, Graves M, Sorenson EJ, Barohn RJ, Belsh JM, Lou JS, Levine T, Saperstein D, Miller RG, Scelsa SN; Combination Drug Selection Trial Study Group. A novel, efficient, randomized selection trial comparing combinations of drug therapy for ALS. Amyotroph Lateral Scler. 2008 Aug;9(4):212-22. doi: 10.1080/17482960802195632. PMID 18608093
- [Background] Sniehotta FF. Towards a theory of intentional behaviour change: plans, planning, and self-regulation. Br J Health Psychol. 2009 May;14(Pt 2):261-73. doi: 10.1348/135910708X389042. Epub 2008 Dec 19. PMID 19102817
- [Background] Locke EA, Latham GP. Building a practically useful theory of goal setting and task motivation. A 35-year odyssey. Am Psychol. 2002 Sep;57(9):705-17. doi: 10.1037//0003-066x.57.9.705. PMID 12237980
- [Background] Michie S, Johnston M, Francis J, Hardeman W, Eccles M. From theory to intervention: Mapping theoretically derived behavioural determinants to behaviour change techniques. Applied psychology. 2008;57:660-680.
- [Background] Williams SL, French DP. What are the most effective intervention techniques for changing physical activity self-efficacy and physical activity behaviour--and are they the same? Health Educ Res. 2011 Apr;26(2):308-22. doi: 10.1093/her/cyr005. Epub 2011 Feb 14. PMID 21321008
- [Background] Mander AP, Sweeting MJ. A product of independent beta probabilities dose escalation design for dual-agent phase I trials. Stat Med. 2015 Apr 15;34(8):1261-76. doi: 10.1002/sim.6434. Epub 2015 Jan 29. PMID 25630638
- [Background] Oe Y, Shimbo D, Ishikawa J, Okajima K, Hasegawa T, Diaz KM, Muntner P, Homma S, Schwartz JE. Alterations in diastolic function in masked hypertension: findings from the masked hypertension study. Am J Hypertens. 2013 Jun;26(6):808-15. doi: 10.1093/ajh/hpt021. Epub 2013 Feb 27. PMID 23446956
- [Background] Booth JN 3rd, Muntner P, Diaz KM, Viera AJ, Bello NA, Schwartz JE, Shimbo D. Evaluation of Criteria to Detect Masked Hypertension. J Clin Hypertens (Greenwich). 2016 Nov;18(11):1086-1094. doi: 10.1111/jch.12830. Epub 2016 Apr 29. PMID 27126770
- [Background] Ensari I, Burg MM, Diaz KM, Fu J, Duran AT, Suls JM, Sumner JA, Monane R, Julian JE, Zhao S, Chaplin WF, Shimbo D. Putative mechanisms Underlying Myocardial infarction onset and Emotions (PUME): a randomised controlled study protocol. BMJ Open. 2018 May 31;8(5):e020525. doi: 10.1136/bmjopen-2017-020525. PMID 29858417
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] Muntner P, Einhorn PT, Cushman WC, Whelton PK, Bello NA, Drawz PE, Green BB, Jones DW, Juraschek SP, Margolis KL, Miller ER 3rd, Navar AM, Ostchega Y, Rakotz MK, Rosner B, Schwartz JE, Shimbo D, Stergiou GS, Townsend RR, Williamson JD, Wright JT Jr, Appel LJ; 2017 National Heart, Lung, and Blood Institute Working Group. Blood Pressure Assessment in Adults in Clinical Practice and Clinic-Based Research: JACC Scientific Expert Panel. J Am Coll Cardiol. 2019 Jan 29;73(3):317-335. doi: 10.1016/j.jacc.2018.10.069. PMID 30678763
- [Background] Schwartz JE, Burg MM, Shimbo D, Broderick JE, Stone AA, Ishikawa J, Sloan R, Yurgel T, Grossman S, Pickering TG. Clinic Blood Pressure Underestimates Ambulatory Blood Pressure in an Untreated Employer-Based US Population: Results From the Masked Hypertension Study. Circulation. 2016 Dec 6;134(23):1794-1807. doi: 10.1161/CIRCULATIONAHA.116.023404. PMID 27920072
- [Background] Anstey DE, Muntner P, Bello NA, Pugliese DN, Yano Y, Kronish IM, Reynolds K, Schwartz JE, Shimbo D. Diagnosing Masked Hypertension Using Ambulatory Blood Pressure Monitoring, Home Blood Pressure Monitoring, or Both? Hypertension. 2018 Nov;72(5):1200-1207. doi: 10.1161/HYPERTENSIONAHA.118.11319. PMID 30354812
- [Background] Reyes-Soffer G, Ngai CI, Lovato L, Karmally W, Ramakrishnan R, Holleran S, Ginsberg HN. Effect of combination therapy with fenofibrate and simvastatin on postprandial lipemia in the ACCORD lipid trial. Diabetes Care. 2013 Feb;36(2):422-8. doi: 10.2337/dc11-2556. Epub 2012 Oct 1. PMID 23033246
- [Background] Reyes G, Yasunaga K, Rothenstein E, Karmally W, Ramakrishnan R, Holleran S, Ginsberg HN. Effects of a 1,3-diacylglycerol oil-enriched diet on postprandial lipemia in people with insulin resistance. J Lipid Res. 2008 Mar;49(3):670-8. doi: 10.1194/jlr.P700019-JLR200. Epub 2007 Dec 18. PMID 18089891
- [Background] Davidson MH, Stein EA, Bays HE, Maki KC, Doyle RT, Shalwitz RA, Ballantyne CM, Ginsberg HN; COMBination of prescription Omega-3 with Simvastatin (COMBOS) Investigators. Efficacy and tolerability of adding prescription omega-3 fatty acids 4 g/d to simvastatin 40 mg/d in hypertriglyceridemic patients: an 8-week, randomized, double-blind, placebo-controlled study. Clin Ther. 2007 Jul;29(7):1354-67. doi: 10.1016/j.clinthera.2007.07.018. PMID 17825687
- [Background] ACCORD Study Group; Buse JB, Bigger JT, Byington RP, Cooper LS, Cushman WC, Friedewald WT, Genuth S, Gerstein HC, Ginsberg HN, Goff DC Jr, Grimm RH Jr, Margolis KL, Probstfield JL, Simons-Morton DG, Sullivan MD. Action to Control Cardiovascular Risk in Diabetes (ACCORD) trial: design and methods. Am J Cardiol. 2007 Jun 18;99(12A):21i-33i. doi: 10.1016/j.amjcard.2007.03.003. Epub 2007 Apr 16. PMID 17599422
- [Background] Karmally W, Montez MG, Palmas W, Martinez W, Branstetter A, Ramakrishnan R, Holleran SF, Haffner SM, Ginsberg HN. Cholesterol-lowering benefits of oat-containing cereal in Hispanic americans. J Am Diet Assoc. 2005 Jun;105(6):967-70. doi: 10.1016/j.jada.2005.03.006. PMID 15942550
- [Background] Kastelein JJ, Ginsberg HN, Langslet G, Hovingh GK, Ceska R, Dufour R, Blom D, Civeira F, Krempf M, Lorenzato C, Zhao J, Pordy R, Baccara-Dinet MT, Gipe DA, Geiger MJ, Farnier M. ODYSSEY FH I and FH II: 78 week results with alirocumab treatment in 735 patients with heterozygous familial hypercholesterolaemia. Eur Heart J. 2015 Nov 14;36(43):2996-3003. doi: 10.1093/eurheartj/ehv370. Epub 2015 Sep 1. PMID 26330422
- [Background] Ginsberg HN, Barr SL, Gilbert A, Karmally W, Deckelbaum R, Kaplan K, Ramakrishnan R, Holleran S, Dell RB. Reduction of plasma cholesterol levels in normal men on an American Heart Association Step 1 diet or a Step 1 diet with added monounsaturated fat. N Engl J Med. 1990 Mar 1;322(9):574-9. doi: 10.1056/NEJM199003013220902. PMID 2304504
- [Background] Nagashima K, Lopez C, Donovan D, Ngai C, Fontanez N, Bensadoun A, Fruchart-Najib J, Holleran S, Cohn JS, Ramakrishnan R, Ginsberg HN. Effects of the PPARgamma agonist pioglitazone on lipoprotein metabolism in patients with type 2 diabetes mellitus. J Clin Invest. 2005 May;115(5):1323-32. doi: 10.1172/JCI23219. Epub 2005 Apr 1. PMID 15841215
- [Background] Ginsberg HN, Karmally W, Siddiqui M, Holleran S, Tall AR, Rumsey SC, Deckelbaum RJ, Blaner WS, Ramakrishnan R. A dose-response study of the effects of dietary cholesterol on fasting and postprandial lipid and lipoprotein metabolism in healthy young men. Arterioscler Thromb. 1994 Apr;14(4):576-86. doi: 10.1161/01.atv.14.4.576. PMID 8148356
- [Background] Saland JM, Satlin LM, Zalsos-Johnson J, Cremers S, Ginsberg HN. Impaired postprandial lipemic response in chronic kidney disease. Kidney Int. 2016 Jul;90(1):172-80. doi: 10.1016/j.kint.2016.02.031. Epub 2016 May 7. PMID 27162092
- [Background] Ginsberg HN, Kris-Etherton P, Dennis B, Elmer PJ, Ershow A, Lefevre M, Pearson T, Roheim P, Ramakrishnan R, Reed R, Stewart K, Stewart P, Phillips K, Anderson N. Effects of reducing dietary saturated fatty acids on plasma lipids and lipoproteins in healthy subjects: the DELTA Study, protocol 1. Arterioscler Thromb Vasc Biol. 1998 Mar;18(3):441-9. doi: 10.1161/01.atv.18.3.441. PMID 9514413
- [Background] Fard A, Tuck CH, Donis JA, Sciacca R, Di Tullio MR, Wu HD, Bryant TA, Chen NT, Torres-Tamayo M, Ramasamy R, Berglund L, Ginsberg HN, Homma S, Cannon PJ. Acute elevations of plasma asymmetric dimethylarginine and impaired endothelial function in response to a high-fat meal in patients with type 2 diabetes. Arterioscler Thromb Vasc Biol. 2000 Sep;20(9):2039-44. doi: 10.1161/01.atv.20.9.2039. PMID 10978246
- [Background] Berglund L, Lefevre M, Ginsberg HN, Kris-Etherton PM, Elmer PJ, Stewart PW, Ershow A, Pearson TA, Dennis BH, Roheim PS, Ramakrishnan R, Reed R, Stewart K, Phillips KM; DELTA Investigators. Comparison of monounsaturated fat with carbohydrates as a replacement for saturated fat in subjects with a high metabolic risk profile: studies in the fasting and postprandial states. Am J Clin Nutr. 2007 Dec;86(6):1611-20. doi: 10.1093/ajcn/86.5.1611. PMID 18065577
- [Background] Ginsberg HN, Jones J, Blaner WS, Thomas A, Karmally W, Fields L, Blood D, Begg MD. Association of postprandial triglyceride and retinyl palmitate responses with newly diagnosed exercise-induced myocardial ischemia in middle-aged men and women. Arterioscler Thromb Vasc Biol. 1995 Nov;15(11):1829-38. doi: 10.1161/01.atv.15.11.1829. PMID 7583562
- [Background] Cheung YK. Sample size formulae for the Bayesian continual reassessment method. Clin Trials. 2013;10(6):852-61. doi: 10.1177/1740774513497294. Epub 2013 Aug 21. PMID 23965547
- [Background] Cheung YK. Coherence principles in dose-finding studies. Biometrika. 2005;92:863-873.
- [Background] Cheung YK. Dose finding by the continual reassessment method. Boca Raton: Taylor & Francis; 2011.
- [Background] Lee SM, Ying Kuen Cheung. Model calibration in the continual reassessment method. Clin Trials. 2009 Jun;6(3):227-38. doi: 10.1177/1740774509105076. PMID 19528132
- [Background] Lee SM, Cheung YK. Calibration of prior variance in the Bayesian continual reassessment method. Stat Med. 2011 Jul 30;30(17):2081-9. doi: 10.1002/sim.4139. Epub 2011 Mar 17. PMID 21413054
- [Background] Wheeler GM, Sweeting MJ, Mander AP, Lee SM, Cheung YK. Modelling semi-attributable toxicity in dual-agent phase I trials with non-concurrent drug administration. Stat Med. 2017 Jan 30;36(2):225-241. doi: 10.1002/sim.6912. Epub 2016 Feb 19. PMID 26891942
- [Background] Cheung YK, Chakraborty B, Davidson KW. Sequential multiple assignment randomized trial (SMART) with adaptive randomization for quality improvement in depression treatment program. Biometrics. 2015 Jun;71(2):450-9. doi: 10.1111/biom.12258. Epub 2014 Oct 29. PMID 25354029
- [Background] Li Y, Wang M, Cheung YK. Treatment and dose prioritization in early phase platform trials of targeted cancer therapies. Journal of the Royal Statistical Society: Series C (Applied Statistics). 2019;68:475-491.
- [Background] Berry DA, Eick SG. Adaptive assignment versus balanced randomization in clinical trials: a decision analysis. Stat Med. 1995 Feb 15;14(3):231-46. doi: 10.1002/sim.4780140302. PMID 7724909
- [Background] Cheung YK, Inoue LY, Wathen JK, Thall PF. Continuous Bayesian adaptive randomization based on event times with covariates. Stat Med. 2006 Jan 15;25(1):55-70. doi: 10.1002/sim.2247. PMID 16025549
- [Background] Wei L, Durham S. The randomized play-the-winner rule in medical trials. Journal of the American Statistical Association. 1978;73:840-843.
- [Background] Kadane JB. Bayesian methods and ethics in a clinical trial design. John Wiley & Sons; 2011.
- [Background] Abel MG, Hannon JC, Sell K, Lillie T, Conlin G, Anderson D. Validation of the Kenz Lifecorder EX and ActiGraph GT1M accelerometers for walking and running in adults. Appl Physiol Nutr Metab. 2008 Dec;33(6):1155-64. doi: 10.1139/h08-103. PMID 19088773
- [Background] Aguilar-Farias N, Brown WJ, Peeters GM. ActiGraph GT3X+ cut-points for identifying sedentary behaviour in older adults in free-living environments. J Sci Med Sport. 2014 May;17(3):293-9. doi: 10.1016/j.jsams.2013.07.002. Epub 2013 Aug 8. PMID 23932934
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Hendelman D, Miller K, Baggett C, Debold E, Freedson P. Validity of accelerometry for the assessment of moderate intensity physical activity in the field. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S442-9. doi: 10.1097/00005768-200009001-00002. PMID 10993413
- [Background] Koster A, Shiroma EJ, Caserotti P, Matthews CE, Chen KY, Glynn NW, Harris TB. Comparison of Sedentary Estimates between activPAL and Hip- and Wrist-Worn ActiGraph. Med Sci Sports Exerc. 2016 Aug;48(8):1514-1522. doi: 10.1249/MSS.0000000000000924. PMID 27031744
- [Background] Plasqui G, Westerterp KR. Physical activity assessment with accelerometers: an evaluation against doubly labeled water. Obesity (Silver Spring). 2007 Oct;15(10):2371-9. doi: 10.1038/oby.2007.281. PMID 17925461
- [Background] Rowlands AV, Thomas PW, Eston RG, Topping R. Validation of the RT3 triaxial accelerometer for the assessment of physical activity. Med Sci Sports Exerc. 2004 Mar;36(3):518-24. doi: 10.1249/01.mss.0000117158.14542.e7. PMID 15076796
- [Background] Van Domelen DR. Accelerometry: Functions for Processing Accelerometer Data. 2018. R package version. 2018 Aug 23;3(2).
- [Background] Schofield WN. Predicting basal metabolic rate, new standards and review of previous work. Hum Nutr Clin Nutr. 1985;39 Suppl 1:5-41. PMID 4044297
- [Background] Dempsey PC, Larsen RN, Sethi P, Sacre JW, Straznicky NE, Cohen ND, Cerin E, Lambert GW, Owen N, Kingwell BA, Dunstan DW. Benefits for Type 2 Diabetes of Interrupting Prolonged Sitting With Brief Bouts of Light Walking or Simple Resistance Activities. Diabetes Care. 2016 Jun;39(6):964-72. doi: 10.2337/dc15-2336. Epub 2016 Apr 13. PMID 27208318
- [Background] Dempsey PC, Sacre JW, Larsen RN, Straznicky NE, Sethi P, Cohen ND, Cerin E, Lambert GW, Owen N, Kingwell BA, Dunstan DW. Interrupting prolonged sitting with brief bouts of light walking or simple resistance activities reduces resting blood pressure and plasma noradrenaline in type 2 diabetes. J Hypertens. 2016 Dec;34(12):2376-2382. doi: 10.1097/HJH.0000000000001101. PMID 27512975
- [Background] Lee IM, Buchner DM. The importance of walking to public health. Med Sci Sports Exerc. 2008 Jul;40(7 Suppl):S512-8. doi: 10.1249/MSS.0b013e31817c65d0. PMID 18562968
- [Background] Morris JN, Hardman AE. Walking to health. Sports Med. 1997 May;23(5):306-32. doi: 10.2165/00007256-199723050-00004. PMID 9181668
- [Background] Mikines KJ, Sonne B, Farrell PA, Tronier B, Galbo H. Effect of physical exercise on sensitivity and responsiveness to insulin in humans. Am J Physiol. 1988 Mar;254(3 Pt 1):E248-59. doi: 10.1152/ajpendo.1988.254.3.E248. PMID 3126668
- [Background] Hamer M. The anti-hypertensive effects of exercise: integrating acute and chronic mechanisms. Sports Med. 2006;36(2):109-16. doi: 10.2165/00007256-200636020-00002. PMID 16464120
- [Background] Carter S, Hartman Y, Holder S, Thijssen DH, Hopkins ND. Sedentary Behavior and Cardiovascular Disease Risk: Mediating Mechanisms. Exerc Sport Sci Rev. 2017 Apr;45(2):80-86. doi: 10.1249/JES.0000000000000106. PMID 28118158
- [Background] Dempsey PC, Larsen RN, Dunstan DW, Owen N, Kingwell BA. Sitting Less and Moving More: Implications for Hypertension. Hypertension. 2018 Nov;72(5):1037-1046. doi: 10.1161/HYPERTENSIONAHA.118.11190. No abstract available. PMID 30354827
- [Background] Peddie MC, Rehrer NJ, Perry TL. Physical activity and postprandial lipidemia: are energy expenditure and lipoprotein lipase activity the real modulators of the positive effect? Prog Lipid Res. 2012 Jan;51(1):11-22. doi: 10.1016/j.plipres.2011.11.002. Epub 2011 Nov 19. PMID 22123195
- [Background] Shvartz E, Gaume JG, White RT, Reibold RC. Hemodynamic responses during prolonged sitting. J Appl Physiol Respir Environ Exerc Physiol. 1983 Jun;54(6):1673-80. doi: 10.1152/jappl.1983.54.6.1673. PMID 6874492
- [Background] Padilla J, Sheldon RD, Sitar DM, Newcomer SC. Impact of acute exposure to increased hydrostatic pressure and reduced shear rate on conduit artery endothelial function: a limb-specific response. Am J Physiol Heart Circ Physiol. 2009 Sep;297(3):H1103-8. doi: 10.1152/ajpheart.00167.2009. Epub 2009 Jul 24. PMID 19633210
- [Background] Padilla J, Fadel PJ. Prolonged sitting leg vasculopathy: contributing factors and clinical implications. Am J Physiol Heart Circ Physiol. 2017 Oct 1;313(4):H722-H728. doi: 10.1152/ajpheart.00326.2017. Epub 2017 Jul 21. PMID 28733451
- [Background] Winkel J, Jorgensen K. Evaluation of foot swelling and lower-limb temperatures in relation to leg activity during long-term seated office work. Ergonomics. 1986 Feb;29(2):313-28. doi: 10.1080/00140138608968267. No abstract available. PMID 3514205
- [Background] Pottier M, Dubreuil A, Monod H. The effects of sitting posture on the volume of the foot. Ergonomics. 1969 Sep;12(5):753-8. doi: 10.1080/00140136908931092. No abstract available. PMID 5361453
- [Background] Mittermayr M, Fries D, Gruber H, Peer S, Klingler A, Fischbach U, Gunga HC, Koralewski E, Faulhaber M, Simmer M, Schobersberger W. Leg edema formation and venous blood flow velocity during a simulated long-haul flight. Thromb Res. 2007;120(4):497-504. doi: 10.1016/j.thromres.2006.12.012. Epub 2007 Jan 23. PMID 17250877
- [Background] Thosar SS, Johnson BD, Johnston JD, Wallace JP. Sitting and endothelial dysfunction: the role of shear stress. Med Sci Monit. 2012 Dec;18(12):RA173-80. doi: 10.12659/msm.883589. PMID 23197245
- [Background] Guo C, Zhou Q, Zhang D, Qin P, Li Q, Tian G, Liu D, Chen X, Liu L, Liu F, Cheng C, Qie R, Han M, Huang S, Wu X, Zhao Y, Ren Y, Zhang M, Liu Y, Hu D. Association of total sedentary behaviour and television viewing with risk of overweight/obesity, type 2 diabetes and hypertension: A dose-response meta-analysis. Diabetes Obes Metab. 2020 Jan;22(1):79-90. doi: 10.1111/dom.13867. Epub 2019 Oct 1. PMID 31468597
- [Background] O'Brien E, Mee F, Atkins N, O'Malley K. Accuracy of the SpaceLabs 90207 determined by the British Hypertension Society protocol. J Hypertens. 1991 Jun;9(6):573-4. doi: 10.1097/00004872-199106000-00016. No abstract available. PMID 1653299
- [Background] Baumgart P, Kamp J. Accuracy of the SpaceLabs Medical 90217 ambulatory blood pressure monitor. Blood Press Monit. 1998 Oct;3(5):303-307. PMID 10212370
- [Background] Groppelli A, Omboni S, Ravogli A, Villani A, Parati G, Mancia G. Validation of the SpaceLabs 90202 and 90207 devices for ambulatory blood pressure monitoring by comparison with intra-arterial resting and ambulatory measurements. J Hypertens Suppl. 1991 Dec;9(6):S334-5. No abstract available. PMID 1818988
- [Background] Diaz KM, Veerabhadrappa P, Kashem MA, Feairheller DL, Sturgeon KM, Williamson ST, Crabbe DL, Brown MD. Relationship of visit-to-visit and ambulatory blood pressure variability to vascular function in African Americans. Hypertens Res. 2012 Jan;35(1):55-61. doi: 10.1038/hr.2011.135. Epub 2011 Aug 4. PMID 21814215
- [Background] Dabl Educational Trust. Sphygmomanometers for ambulatory blood pressure measurement. 2014; http://www.dableducational.org/sphygmomanometers/devices_3_abpm.html Accessed October 1, 2019.
- [Background] Krause T, Lovibond K, Caulfield M, McCormack T, Williams B; Guideline Development Group. Management of hypertension: summary of NICE guidance. BMJ. 2011 Aug 25;343:d4891. doi: 10.1136/bmj.d4891. No abstract available. PMID 21868454
- [Background] Richter EA, Hargreaves M. Exercise, GLUT4, and skeletal muscle glucose uptake. Physiol Rev. 2013 Jul;93(3):993-1017. doi: 10.1152/physrev.00038.2012. PMID 23899560
- [Background] Hamilton MT, Hamilton DG, Zderic TW. Role of low energy expenditure and sitting in obesity, metabolic syndrome, type 2 diabetes, and cardiovascular disease. Diabetes. 2007 Nov;56(11):2655-67. doi: 10.2337/db07-0882. Epub 2007 Sep 7. PMID 17827399
- [Background] Hamilton MT, Hamilton DG, Zderic TW. The Necessity of Active Muscle Metabolism for Healthy Aging: Muscular Activity Throughout the Entire Day. Prog Mol Biol Transl Sci. 2018;155:53-68. doi: 10.1016/bs.pmbts.2017.12.014. Epub 2018 Feb 24. PMID 29653682
- [Background] Dempsey PC, Owen N, Yates TE, Kingwell BA, Dunstan DW. Sitting Less and Moving More: Improved Glycaemic Control for Type 2 Diabetes Prevention and Management. Curr Diab Rep. 2016 Nov;16(11):114. doi: 10.1007/s11892-016-0797-4. PMID 27699700
- [Background] Loh R, Stamatakis E, Folkerts D, Allgrove JE, Moir HJ. Effects of Interrupting Prolonged Sitting with Physical Activity Breaks on Blood Glucose, Insulin and Triacylglycerol Measures: A Systematic Review and Meta-analysis. Sports Med. 2020 Feb;50(2):295-330. doi: 10.1007/s40279-019-01183-w. PMID 31552570
- [Background] Powell C, Herring MP, Dowd KP, Donnelly AE, Carson BP. The cross-sectional associations between objectively measured sedentary time and cardiometabolic health markers in adults - a systematic review with meta-analysis component. Obes Rev. 2018 Mar;19(3):381-395. doi: 10.1111/obr.12642. Epub 2017 Nov 27. PMID 29178252
- [Background] Wu AHB. Tietz clinical guide to laboratory tests. St. Louis, Mo.: Saunders/Elsevier; 2006.
- [Background] Allison DB, Paultre F, Maggio C, Mezzitis N, Pi-Sunyer FX. The use of areas under curves in diabetes research. Diabetes Care. 1995 Feb;18(2):245-50. doi: 10.2337/diacare.18.2.245. PMID 7729306
- [Background] Voils CI, King HA, Maciejewski ML, Allen KD, Yancy WS Jr, Shaffer JA. Approaches for informing optimal dose of behavioral interventions. Ann Behav Med. 2014 Dec;48(3):392-401. doi: 10.1007/s12160-014-9618-7. PMID 24722964
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Gauvin L, Rejeski WJ. The exercise-induced feeling inventory: Development and initial validation. Journal of Sport and Exercise Psychology. 1993;15:403-423.
- [Background] Focht BC, Knapp DJ, Gavin TP, Raedeke TD, Hickner RC. Affective and self-efficacy responses to acute aerobic exercise in sedentary older and younger adults. J Aging Phys Act. 2007 Apr;15(2):123-38. doi: 10.1123/japa.15.2.123. PMID 17556780
- [Background] Focht BC. Brief walks in outdoor and laboratory environments: effects on affective responses, enjoyment, and intentions to walk for exercise. Res Q Exerc Sport. 2009 Sep;80(3):611-20. doi: 10.1080/02701367.2009.10599600. PMID 19791648
- [Background] Annesi JJ. Relationship between before-to-after-exercise feeling state changes and exercise session attendance over 14 weeks: Testing principles of operant conditioning. European Journal of Sport Science. 2005;5:159-163.
- [Background] Williams DM. Psychological hedonism, hedonic motivation, and health behavior. Affective determinants of health behavior. 2018:204.
- [Background] Williams DM, Dunsiger S, Ciccolo JT, Lewis BA, Albrecht AE, Marcus BH. Acute Affective Response to a Moderate-intensity Exercise Stimulus Predicts Physical Activity Participation 6 and 12 Months Later. Psychol Sport Exerc. 2008 May;9(3):231-245. doi: 10.1016/j.psychsport.2007.04.002. No abstract available. PMID 18496608
- [Background] Bryan A, Hutchison KE, Seals DR, Allen DL. A transdisciplinary model integrating genetic, physiological, and psychological correlates of voluntary exercise. Health Psychol. 2007 Jan;26(1):30-9. doi: 10.1037/0278-6133.26.1.30. PMID 17209695
- [Background] Williams DM. Exercise, affect, and adherence: an integrated model and a case for self-paced exercise. J Sport Exerc Psychol. 2008 Oct;30(5):471-96. doi: 10.1123/jsep.30.5.471. PMID 18971508
- [Background] Ekkekakis P. Pleasure and displeasure from the body: Perspectives from exercise. Cogn Emot. 2003 Mar;17(2):213-239. doi: 10.1080/02699930302292. PMID 29715726
- [Background] Ekkekakis P, Petruzzello SJ. Analysis of the affect measurement conundrum in exercise psychology: IV. A conceptual case for the affect circumplex. Psychology of Sport and Exercise. 2002;3:35-63.
- [Background] Hardy CJ, Rejeski WJ. Not what, but how one feels: The measurement of affect during exercise. Journal of sport and exercise psychology. 1989;11:304-317.
- [Background] Williams DM, Dunsiger S, Jennings EG, Marcus BH. Does affective valence during and immediately following a 10-min walk predict concurrent and future physical activity? Ann Behav Med. 2012 Aug;44(1):43-51. doi: 10.1007/s12160-012-9362-9. PMID 22532005
- [Background] Rhodes RE, Kates A. Can the Affective Response to Exercise Predict Future Motives and Physical Activity Behavior? A Systematic Review of Published Evidence. Ann Behav Med. 2015 Oct;49(5):715-31. doi: 10.1007/s12160-015-9704-5. PMID 25921307
- [Background] Mongey S, Pilossoph L, Weinberg A. Which workers bear the burden of social distancing? J Econ Inequal. 2021;19(3):509-526. doi: 10.1007/s10888-021-09487-6. Epub 2021 Aug 2. PMID 34366750
- [Background] Schaufeli WB, Bakker AB, Salanova M. The measurement of work engagement with a short questionnaire - A cross-national study. Educ Psychol Meas. 2006;66:701-716.
- [Background] Bryan J, Tuckey M, Einother SJ, Garczarek U, Garrick A, De Bruin EA. Relationships between tea and other beverage consumption to work performance and mood. Appetite. 2012 Feb;58(1):339-46. doi: 10.1016/j.appet.2011.11.009. Epub 2011 Nov 12. PMID 22100487
- [Background] Lanaj K, Johnson RE, Barnes CM. Beginning the workday yet already depleted? Consequences of late-night smartphone use and sleep. Organ Behav Hum Dec. 2014;124:11-23.
- [Background] Seppala P, Mauno S, Feldt T, Hakanen J, Kinnunen U, Tolvanen A, Schaufeli W. The Construct Validity of the Utrecht Work Engagement Scale: Multisample and Longitudinal Evidence. J Happiness Stud. 2009;10:459-481.
- [Background] Kessler RC, Barber C, Beck A, Berglund P, Cleary PD, McKenas D, Pronk N, Simon G, Stang P, Ustun TB, Wang P. The World Health Organization Health and Work Performance Questionnaire (HPQ). J Occup Environ Med. 2003 Feb;45(2):156-74. doi: 10.1097/01.jom.0000052967.43131.51. PMID 12625231
- [Background] World Health Organization. Waist circumference and waist-hip ratio: Report of a WHO expert consultation. Geneva, Switzerland: World Health Organization; 2008.
- [Background] Cornelissen VA, Smart NA. Exercise training for blood pressure: a systematic review and meta-analysis. J Am Heart Assoc. 2013 Feb 1;2(1):e004473. doi: 10.1161/JAHA.112.004473. PMID 23525435
- [Background] Cornelissen VA, Buys R, Smart NA. Endurance exercise beneficially affects ambulatory blood pressure: a systematic review and meta-analysis. J Hypertens. 2013 Apr;31(4):639-48. doi: 10.1097/HJH.0b013e32835ca964. PMID 23325392
- [Background] Pescatello LS, Kulikowich JM. The aftereffects of dynamic exercise on ambulatory blood pressure. Med Sci Sports Exerc. 2001 Nov;33(11):1855-61. doi: 10.1097/00005768-200111000-00009. PMID 11689735
- [Background] Cardoso CG Jr, Gomides RS, Queiroz AC, Pinto LG, da Silveira Lobo F, Tinucci T, Mion D Jr, de Moraes Forjaz CL. Acute and chronic effects of aerobic and resistance exercise on ambulatory blood pressure. Clinics (Sao Paulo). 2010 Mar;65(3):317-25. doi: 10.1590/S1807-59322010000300013. PMID 20360924
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Eckel RH, Jakicic JM, Ard JD, de Jesus JM, Houston Miller N, Hubbard VS, Lee IM, Lichtenstein AH, Loria CM, Millen BE, Nonas CA, Sacks FM, Smith SC Jr, Svetkey LP, Wadden TA, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 AHA/ACC guideline on lifestyle management to reduce cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2960-84. doi: 10.1016/j.jacc.2013.11.003. Epub 2013 Nov 12. No abstract available. PMID 24239922
- [Background] Pescatello LS, Franklin BA, Fagard R, Farquhar WB, Kelley GA, Ray CA; American College of Sports Medicine. American College of Sports Medicine position stand. Exercise and hypertension. Med Sci Sports Exerc. 2004 Mar;36(3):533-53. doi: 10.1249/01.mss.0000115224.88514.3a. PMID 15076798
- [Background] Law MR, Morris JK, Wald NJ. Use of blood pressure lowering drugs in the prevention of cardiovascular disease: meta-analysis of 147 randomised trials in the context of expectations from prospective epidemiological studies. BMJ. 2009 May 19;338:b1665. doi: 10.1136/bmj.b1665. PMID 19454737
- [Background] Oberlin DJ, Mikus CR, Kearney ML, Hinton PS, Manrique C, Leidy HJ, Kanaley JA, Rector RS, Thyfault JP. One bout of exercise alters free-living postprandial glycemia in type 2 diabetes. Med Sci Sports Exerc. 2014 Feb;46(2):232-8. doi: 10.1249/MSS.0b013e3182a54d85. PMID 23872939
- [Background] Rynders CA, Weltman JY, Jiang B, Breton M, Patrie J, Barrett EJ, Weltman A. Effects of exercise intensity on postprandial improvement in glucose disposal and insulin sensitivity in prediabetic adults. J Clin Endocrinol Metab. 2014 Jan;99(1):220-8. doi: 10.1210/jc.2013-2687. Epub 2013 Dec 20. PMID 24243632
- [Background] Ross R, Dagnone D, Jones PJ, Smith H, Paddags A, Hudson R, Janssen I. Reduction in obesity and related comorbid conditions after diet-induced weight loss or exercise-induced weight loss in men. A randomized, controlled trial. Ann Intern Med. 2000 Jul 18;133(2):92-103. doi: 10.7326/0003-4819-133-2-200007180-00008. PMID 10896648
- [Background] Weiss EP, Racette SB, Villareal DT, Fontana L, Steger-May K, Schechtman KB, Klein S, Holloszy JO; Washington University School of Medicine CALERIE Group. Improvements in glucose tolerance and insulin action induced by increasing energy expenditure or decreasing energy intake: a randomized controlled trial. Am J Clin Nutr. 2006 Nov;84(5):1033-42. doi: 10.1093/ajcn/84.5.1033. PMID 17093155
- [Background] Bouchonville M, Armamento-Villareal R, Shah K, Napoli N, Sinacore DR, Qualls C, Villareal DT. Weight loss, exercise or both and cardiometabolic risk factors in obese older adults: results of a randomized controlled trial. Int J Obes (Lond). 2014 Mar;38(3):423-31. doi: 10.1038/ijo.2013.122. Epub 2013 Jul 4. PMID 23823329
- [Background] Alyass A, Almgren P, Akerlund M, Dushoff J, Isomaa B, Nilsson P, Tuomi T, Lyssenko V, Groop L, Meyre D. Modelling of OGTT curve identifies 1 h plasma glucose level as a strong predictor of incident type 2 diabetes: results from two prospective cohorts. Diabetologia. 2015 Jan;58(1):87-97. doi: 10.1007/s00125-014-3390-x. Epub 2014 Oct 8. PMID 25292440
- [Background] Feizi A, Meamar R, Eslamian M, Amini M, Nasri M, Iraj B. Area under the curve during OGTT in first-degree relatives of diabetic patients as an efficient indicator of future risk of type 2 diabetes and prediabetes. Clin Endocrinol (Oxf). 2017 Dec;87(6):696-705. doi: 10.1111/cen.13443. Epub 2017 Sep 20. PMID 28793372
- [Background] Cheung YK, Chappell R. Sequential designs for phase I clinical trials with late-onset toxicities. Biometrics. 2000 Dec;56(4):1177-82. doi: 10.1111/j.0006-341x.2000.01177.x. PMID 11129476
- [Background] Cheung YK, Thall PF. Monitoring the rates of composite events with censored data in phase II clinical trials. Biometrics. 2002 Mar;58(1):89-97. doi: 10.1111/j.0006-341x.2002.00089.x. PMID 11890331
- [Background] Chastin SFM, De Craemer M, De Cocker K, Powell L, Van Cauwenberg J, Dall P, Hamer M, Stamatakis E. How does light-intensity physical activity associate with adult cardiometabolic health and mortality? Systematic review with meta-analysis of experimental and observational studies. Br J Sports Med. 2019 Mar;53(6):370-376. doi: 10.1136/bjsports-2017-097563. Epub 2018 Apr 25. PMID 29695511
- [Background] Henriksen EJ. Invited review: Effects of acute exercise and exercise training on insulin resistance. J Appl Physiol (1985). 2002 Aug;93(2):788-96. doi: 10.1152/japplphysiol.01219.2001. PMID 12133893
- [Background] Casonatto J, Goessler KF, Cornelissen VA, Cardoso JR, Polito MD. The blood pressure-lowering effect of a single bout of resistance exercise: A systematic review and meta-analysis of randomised controlled trials. Eur J Prev Cardiol. 2016 Nov;23(16):1700-1714. doi: 10.1177/2047487316664147. Epub 2016 Aug 10. PMID 27512052
- [Background] Wong GW, Boyda HN, Wright JM. Blood pressure lowering efficacy of beta-1 selective beta blockers for primary hypertension. Cochrane Database Syst Rev. 2016 Mar 10;3(3):CD007451. doi: 10.1002/14651858.CD007451.pub2. PMID 26961574
- [Background] Brook RD, Appel LJ, Rubenfire M, Ogedegbe G, Bisognano JD, Elliott WJ, Fuchs FD, Hughes JW, Lackland DT, Staffileno BA, Townsend RR, Rajagopalan S; American Heart Association Professional Education Committee of the Council for High Blood Pressure Research, Council on Cardiovascular and Stroke Nursing, Council on Epidemiology and Prevention, and Council on Nutrition, Physical Activity. Beyond medications and diet: alternative approaches to lowering blood pressure: a scientific statement from the american heart association. Hypertension. 2013 Jun;61(6):1360-83. doi: 10.1161/HYP.0b013e318293645f. Epub 2013 Apr 22. PMID 23608661
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force for the Management of Arterial Hypertension of the European Society of Hypertension and the European Society of Cardiology. 2013 ESH/ESC Practice Guidelines for the Management of Arterial Hypertension. Blood Press. 2014 Feb;23(1):3-16. doi: 10.3109/08037051.2014.868629. Epub 2013 Dec 20. No abstract available. PMID 24359485
- [Background] Dasgupta K, Quinn RR, Zarnke KB, Rabi DM, Ravani P, Daskalopoulou SS, Rabkin SW, Trudeau L, Feldman RD, Cloutier L, Prebtani A, Herman RJ, Bacon SL, Gilbert RE, Ruzicka M, McKay DW, Campbell TS, Grover S, Honos G, Schiffrin EL, Bolli P, Wilson TW, Lindsay P, Hill MD, Coutts SB, Gubitz G, Gelfer M, Vallee M, Prasad GV, Lebel M, McLean D, Arnold JM, Moe GW, Howlett JG, Boulanger JM, Larochelle P, Leiter LA, Jones C, Ogilvie RI, Woo V, Kaczorowski J, Burns KD, Petrella RJ, Hiremath S, Milot A, Stone JA, Drouin D, Lavoie KL, Lamarre-Cliche M, Tremblay G, Hamet P, Fodor G, Carruthers SG, Pylypchuk GB, Burgess E, Lewanczuk R, Dresser GK, Penner SB, Hegele RA, McFarlane PA, Khara M, Pipe A, Oh P, Selby P, Sharma M, Reid DJ, Tobe SW, Padwal RS, Poirier L. 2014 canadian hypertension education program recommendations for blood pressure measurement, diagnosis, assessment of risk, prevention, and treatment of hypertension. Can J Cardiol. 2014;30:485-501.
- [Background] Pescatello LS, MacDonald HV, Ash GI, Lamberti LM, Farquhar WB, Arena R, Johnson BT. Assessing the Existing Professional Exercise Recommendations for Hypertension: A Review and Recommendations for Future Research Priorities. Mayo Clin Proc. 2015 Jun;90(6):801-12. doi: 10.1016/j.mayocp.2015.04.008. PMID 26046413
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Tonoli C, Heyman E, Roelands B, Buyse L, Cheung SS, Berthoin S, Meeusen R. Effects of different types of acute and chronic (training) exercise on glycaemic control in type 1 diabetes mellitus: a meta-analysis. Sports Med. 2012 Dec 1;42(12):1059-80. doi: 10.1007/BF03262312. PMID 23134339
- [Background] Liu S, Goodman J, Nolan R, Lacombe S, Thomas SG. Blood pressure responses to acute and chronic exercise are related in prehypertension. Med Sci Sports Exerc. 2012 Sep;44(9):1644-52. doi: 10.1249/MSS.0b013e31825408fb. PMID 22899388
- [Background] Hecksteden A, Grutters T, Meyer T. Associations between acute and chronic effects of exercise on indicators of metabolic health: a pilot training trial. PLoS One. 2013 Nov 21;8(11):e81181. doi: 10.1371/journal.pone.0081181. eCollection 2013. PMID 24278393
- [Background] Haskell WL. J.B. Wolffe Memorial Lecture. Health consequences of physical activity: understanding and challenges regarding dose-response. Med Sci Sports Exerc. 1994 Jun;26(6):649-60. doi: 10.1249/00005768-199406000-00001. PMID 8052103
- [Background] Pescatello LS, MacDonald HV, Lamberti L, Johnson BT. Exercise for Hypertension: A Prescription Update Integrating Existing Recommendations with Emerging Research. Curr Hypertens Rep. 2015 Nov;17(11):87. doi: 10.1007/s11906-015-0600-y. PMID 26423529
- [Background] NIH Human Research Protection Program. Policy and communications Bulletin - The Clinical Center/Medical Administrative Series: Guidelines for Limits of Blood Drawn for Research Purposes in the Clinical Center; 2009. Available at: https://irb.research.chop.edu/sites/default/files/documents/g_nih_blooddraws.pdf.
- [Background] Husain SA, Diaz K, Schwartz JE, Parsons FE, Burg MM, Davidson KW, Kronish IM. Behavioral economics implementation: Regret lottery improves mHealth patient study adherence. Contemp Clin Trials Commun. 2019 May 31;15:100387. doi: 10.1016/j.conctc.2019.100387. eCollection 2019 Sep. PMID 31198881
- [Background] Cheung YK, Hsueh PS, Ensari I, Willey JZ, Diaz KM. Quantile Coarsening Analysis of High-Volume Wearable Activity Data in a Longitudinal Observational Study. Sensors (Basel). 2018 Sep 12;18(9):3056. doi: 10.3390/s18093056. PMID 30213093